CLINICAL TRIAL: NCT04435613
Title: Clinical and Physiological Assessment of a Nearly Ultra-protective Lung Ventilation Strategy: A Quasi-experimental Preliminary Study in ARDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica las Condes, Chile (Other)
Responsible Party: Principal Investigator, Martin Benites, Principal Investigator: Martín Hernán Benites Albanese, Clinica las Condes, Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S022018
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: ARDS; Volumetric Capnography
Keywords: dead space, end-inspiratory pause, respiratory rate, ARDS

STUDY DESIGN:
Intervention Model Description: A quasi-experimental, non-randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- protective mechanical ventilation (Other): Ten patients with moderate to severe ARDS were subjected to a nearly ultra-protective ventilation strategy generating a reduction in minute ventilation (Tidal volume of 5 ml/kg of predicted body weight together with a 20% reduction in respiratory rate). In addition to end-inspiratory pause, prolongation was set to avoid hypercapnia. Protocol phases: Baseline conditions: Tidal volume of 7 ml/kg. I: Tidal volume of 6 ml/kg. II: Tidal volume of 5 ml/kg. III: Increase end-inspiratory pause until achieving an I:E ratio equal to 1. IV: Respiratory rate reduction until 20% of the basal condition keeping constant I:E ratio equal to 1
  Interventions: Other: protective mechanical ventilation strategies

INTERVENTIONS:
Other: protective mechanical ventilation strategies — 1. Reduce tidal volume from 7 ml/kg to 5 ml/kg. 2 Set end-inspiratory pausa. 3 respiratory rate reduction until 20% of the basal condition

SUMMARY:
This study aims to determine whether a protective mechanical ventilator strategy generates a reduction in the Bohr´s dead space in patients with moderate or severe acute respiratory distress syndrome (ARDS). Commonly used ventilatory strategies in the clinical practice were applied sequentially to assess their impact. Data obtained from volumetric capnography will be recorded after each ventilatory strategy is applied

DETAILED DESCRIPTION:
Protective mechanical ventilation strategies are currently the cornerstone of treatment for patients undergoing mechanical ventilatory support. Among them, we can mention the reduction in tidal volume, the reduction in driving pressure, the PEEP setting, and the respiratory rate reduction. All of these strategies are aimed at preventing ventilator-induced lung injury. Few clinical studies have evaluated the effects of protective mechanical ventilation strategies on dead-space. This study was designed to evaluate dead space and alveolar ventilation with a sequence of protective ventilatory strategies, keeping PEEP levels constant. The ventilatory strategy was developed to reduce tidal volume, set an end-inspiratory pause, and reduce the frequencies of lung tissue impact.

Baseline:

All the patients kept the variables under study constant for 60 minutes. Each of the participants was studied for a period of 150 minutes. PEEP programming was set with transpulmonary end-expiratory pressures to maintain between 0 and 5 cmH2O and was remained constant throughout the study.

Protocol design:

Baseline: Vt 7 ml/kg/PBW Phase I: Vt 6 ml/kg/PBW. Phase II: Vt 5 ml/kg/PBW. Phase III: end-inspiratory pause prolongation until achieving I:E ratio equal to 1, maintaining a constant Vt level (5 ml/kg/PBW) Phase IV: Respiratory rate reduction by 20% of basal conditions, maintaining constant VT level (5 ml/kg/PBW).

After 30 minutes of continuous monitoring, minute ventilation, mechanical power, variables obtained by volumetric capnography, and arterial blood gases were recorded in each study phase.

This study will be performed in the Intensive Care Unit of a University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* The requirement of invasive mechanical ventilation for more than 4 hours and less than 72 hours
* Severe hypoxemia (PAFI < 200) secondary to ARDS

Exclusion Criteria:

* Heart failure stage IV
* Chronic obstructive pulmonary disease (COPD) on home oxygen
* Bronchopulmonary fistula
* Hypovolemic Shock with active hemorrhage
* Gastrointestinal bleeding
* Oesophageal Varices
* Nasopharynx surgery, recent oesophageal or gastric surgery
* Massive Pulmonary Thromboembolism
* Catastrophic respiratory failure requiring urgent extracorporeal life support
* Respiratory acidosis. Hydrogen potential (pH) is less than 7.20 and PaCO2 higher than 60 mmHg at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
To analyse the effects of different protective mechanical ventilator strategies on Bohr's dead space (VDBohr/VT) in patients with acute respiratory distress syndrome | 150 minutes
  After the systematic reduction of the tidal volume, end-inspiratory pause prolongation, and the reduction of the respiratory rate, the optimisation of the dead space and the alveolar ventilation could be generated.

CONTACTS AND LOCATIONS:
Overall Officials: Martín Benites Albanese, Physician, Principal Investigator — Critical Care Department, Clínica Las Condes
Locations (1):
- Clínica Las Condes, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Tusman G, Sipmann FS, Borges JB, Hedenstierna G, Bohm SH. Validation of Bohr dead space measured by volumetric capnography. Intensive Care Med. 2011 May;37(5):870-4. doi: 10.1007/s00134-011-2164-x. Epub 2011 Feb 26. PMID 21359609
- [Background] Tusman G, Gogniat E, Bohm SH, Scandurra A, Suarez-Sipmann F, Torroba A, Casella F, Giannasi S, Roman ES. Reference values for volumetric capnography-derived non-invasive parameters in healthy individuals. J Clin Monit Comput. 2013 Jun;27(3):281-8. doi: 10.1007/s10877-013-9433-x. Epub 2013 Feb 7. PMID 23389294
- [Background] Lellouche F, Delorme M, Brochard L. Impact of Respiratory Rate and Dead Space in the Current Era of Lung Protective Mechanical Ventilation. Chest. 2020 Jul;158(1):45-47. doi: 10.1016/j.chest.2020.02.033. Epub 2020 Jul 2. No abstract available. PMID 32654726
- [Background] Astrom E, Uttman L, Niklason L, Aboab J, Brochard L, Jonson B. Pattern of inspiratory gas delivery affects CO2 elimination in health and after acute lung injury. Intensive Care Med. 2008 Feb;34(2):377-84. doi: 10.1007/s00134-007-0840-7. Epub 2007 Sep 1. PMID 17763841
- [Background] Devaquet J, Jonson B, Niklason L, Si Larbi AG, Uttman L, Aboab J, Brochard L. Effects of inspiratory pause on CO2 elimination and arterial PCO2 in acute lung injury. J Appl Physiol (1985). 2008 Dec;105(6):1944-9. doi: 10.1152/japplphysiol.90682.2008. Epub 2008 Sep 18. PMID 18801962
- [Background] Aguirre-Bermeo H, Moran I, Bottiroli M, Italiano S, Parrilla FJ, Plazolles E, Roche-Campo F, Mancebo J. End-inspiratory pause prolongation in acute respiratory distress syndrome patients: effects on gas exchange and mechanics. Ann Intensive Care. 2016 Dec;6(1):81. doi: 10.1186/s13613-016-0183-z. Epub 2016 Aug 24. PMID 27558174

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT04435613/Prot_SAP_000.pdf